CLINICAL TRIAL: NCT02566135
Title: I-gel Versus C-LMA as a Conduit for Tracheal Intubation Using Ventilating Bougie
Brief Title: I-gel Versus Classic-Laryngeal Mask Airway (C-LMA) as a Conduit for Tracheal Intubation Using Ventilating Bougie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College Baroda (Other)
Responsible Party: Principal Investigator, DR ADITI AMRUTLAL DHIMAR, DR ADITI AMRUTLAL DHIMAR, Medical College Baroda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR/85/Inst/GJ/2013
Record Dates: First submitted 2015-09-07; First posted 2015-10-02 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Intubation; Difficult
Keywords: C-LMA; I-gel; ventilating bougie; intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-I (Active Comparator): Tracheal intubation using I-gel and ventilating bougie insertion. In Group-I, following general anaesthesia I-gel is to be inserted, through it ventilating bougie is to be inserted then I-gel is to be removed and endotracheal tube is to be railroaded over ventilating bougie. Then ventilating bougie is to be removed.
  Interventions: Device: Tracheal Intubation using I-gel and ventilating bougie
- Group-C (Active Comparator): Tracheal intubation using C-LMA and ventilating bougie insertion. In Group-C, following general anaesthesia C-LMA is to be inserted, through it ventilating bougie is to be inserted then C-LMA is to be removed and endotracheal tube is to be railroaded over ventilating bougie. Then ventilating bougie is to be removed.
  Interventions: Device: Tracheal Intubation using C-LMA and ventilating bougie

INTERVENTIONS:
Device: Tracheal Intubation using I-gel and ventilating bougie — Following general anaesthesia I-gel was inserted. After proper placement . ventilating bougie was inserted. Once it's placement is confirmed I-gel was removed keeping the ventilating bougie in situ. Then appropriate sized endotracheal tube was railroaded over ventilating bougie then it (v.bouggie) was removed . Proper placement of endotracheal tube was confirmed by bilateral equal chest excursion and air entry on auscultation, absence of gastric insuffflation sound over epigastrium and 'sine' wave on capnography. Maximum 3 attempts were allowed for I-gel, ventilating bougie and endotracheal tube.
  Arms: Group-I
Device: Tracheal Intubation using C-LMA and ventilating bougie — Following general anaesthesia C-LMA was inserted. After proper placement of C-LMA, ventilating bougie was inserted. It's placement was confirmed and C-LMA was removed after deflation of cuff keeping the ventilating bougie in situ. Then appropriate sized endotracheal tube was railroaded over ventilating bougie. It's placement was confirmed by bilateral equal air entry and chest excursion, absence of gastric insufflation sound over epigastrium and 'sine' wave on capnography. Maximum 3 attempts were allowed for C-LMA , ventilating bougie and endotracheal tube.
  Arms: Group-C

SUMMARY:
Supraglottic Airway devices(SGAs) like I-Gel and C-LMA ( classic laryngeal mask airway ) have been used as a conduit for tracheal intubation using ventilating bougie. General Anaesthesia with tracheal intubation is one of the technique for giving anaesthesia. Tracheal intubation may become difficult sometimes and endangers patients life. Using SGAs as a conduit for tracheal intubation helps in securing airway. This will be further facilitated by using ventilating bougie, as it maintains oxygenation.

DETAILED DESCRIPTION:
SGAs have been used as a conduit for tracheal intubation using ventilating bougie. Patients were anaesthetised with intravenous induction agent, non-depolarising muscle relaxant and then SGAs were inserted. Two groups were compared. In group I : I-gel was inserted, its position was confirmed and then ventilating bougie was inserted through it. It's position was confirmed, then I-gel was removed , Endotracheal tube was railroaded over ventilating bougie and it's position was confirmed. In group C : C-LMA was inserted, its position was confirmed and then ventilating bougie was inserted through it. It's position was confirmed, then C-LMA was removed , Endotracheal tube was railroaded over ventilating bougie and it's position was confirmed.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60 years
* Gender : either sex
* American society of Anaesthesiologist's Physical Status (ASAPS) I and II
* Patients posted for surgery requiring general anaesthesia and endotracheal intubation.

Exclusion Criteria:

* age <18 years and > 60 years
* ASAPS III or IV
* Obesity body mass index >25
* Patients with mouth opening <2cms
* Patients with Malampatti grade III and IV
* Patients having history of gastro-esophageal reflux disease
* Patients with history of inadequate fasting
* Patients with known or anticipated difficult tracheal intubation or face-mask ventilation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aditi A Dhimar, M.D.(anaes), Principal Investigator — CDSCO

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapoor S, Jethava DD, Gupta P, Jethava D, Kumar A. Comparison of supraglottic devices i-gel((R)) and LMA Fastrach((R)) as conduit for endotracheal intubation. Indian J Anaesth. 2014 Jul;58(4):397-402. doi: 10.4103/0019-5049.138969. PMID 25197106
- [Result] Wong DT, Yang JJ, Mak HY, Jagannathan N. Use of intubation introducers through a supraglottic airway to facilitate tracheal intubation: a brief review. Can J Anaesth. 2012 Jul;59(7):704-15. doi: 10.1007/s12630-012-9714-8. Epub 2012 Jun 1. PMID 22653838
- [Result] Singh J, Yadav MK, Marahatta SB, Shrestha BL. Randomized crossover comparison of the laryngeal mask airway classic with i-gel laryngeal mask airway in the management of difficult airway in post burn neck contracture patients. Indian J Anaesth. 2012 Jul;56(4):348-52. doi: 10.4103/0019-5049.100815. PMID 23087456

RESULTS

PARTICIPANT FLOW:
Groups:
- Group-I: In Group-I, I-gel is to be used as a conduit for tracheal intubation using ventilating bougie.
  Tracheal Intubation: Following general anaesthesia I-gel was inserted. After proper placement . ventilating bougie was inserted. Once it's placement is confirmed I-gel was removed keeping the ventilating bougie in situ. Then appropriate sized endotracheal tube was railroaded over ventilating bougie then it (v.bouggie) was removed . Proper placement of endotracheal tube was confirmed by bilateral equal chest excursion and air entry on auscultation, absence of gastric insuffflation sound over epigastrium and 'sine' wave on capnography. Maximum 3 attempts were allowed for I-gel, ventilating bougie and endotracheal tube.
- Group-C: In Group-C, C-LMA is to be used as a conduit for tracheal intubation using ventilating bougie.
  Tracheal Intubation: Following general anaesthesia C-LMA was inserted. Aftre proper placement ventilating bougie was inserted. It's placement was confirmed and C-LMA was removed after deflation of cuff keeping the ventilating bougie in situ. Then appropriate sized endotracheal tube was railroaded over ventilating bougie. It's placement was confirmed by bilateral equal air entry and chest excursion, absence of gastric insufflation sound over epigastrium and 'sine' wave on capnography. Maximum 3 attempts were allowed for C-LMA , ventilating bougie and endotracheal tube.
Period: Overall Study
Arm/Group | Group-I | Group-C
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-I | Group-C | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.03 (10.13) | 36.13 (11.24) | 35.58 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 16 | 14 | 30
ASAPS ( American society of Anaesthesiologist's physical ststus [Number; unit: participants] — ASA I:
  A normal healthy patient Healthy, non-smoking, no or minimal alcohol use
  ASA II:
  A patient with mild systemic disease Mild diseases only without substantive functional limitations.
  ASA III:
  A patient with severe systemic disease Substantive functional limitations; One or more moderate to severe diseases.
  ASA IV:
  A patient with severe systemic disease that is a constant threat to life
  ASA V:
  A moribund patient who is not expected to survive without the operation
  ASA VI:
  A declared brain-dead patient whose organs are being removed for donor purposes
  participants
    ASAPS I | 21 | 23 | 44
    ASAPS II | 8 | 6 | 14
BMI (body mass index) [Mean (Standard Deviation); unit: Kg/m2] | 21.30 (2.96) | 21.43 (2.19) | 21.36 (2.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Attempts for I-gel or Classic-LMA Insertions
Time Frame: 60 seconds
Measure: Number; unit: attempt
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
attempt
  1st attempt | 25 | 22
  2nd attempt | 2 | 5
  3rd attempt | 2 | 2
Statistical Analysis 1: Comparison: Group-I vs Group-C; Chi square test was applied to see weather there is a statistical significant difference between group I and group C for attempt for supraglottic airway insertion; Test type: Other; p = 0.5033, Chi-squared, Corrected; Risk Ratio (RR) = 1.4628, 95% CI 2-sided [0.6401 to 3.3428]

2. Primary Outcome: Number of Attempts for Ventilating Bougie Insertions Through I-gel or C-LMA
Time Frame: 45 seconds
Measure: Number; unit: attempt
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
attempt
  1st attempt | 23 | 24
  2nd attempt | 6 | 4
  3rd attempt | 0 | 1
Statistical Analysis 1: Comparison: Group-I vs Group-C; We had applied chi square to see the statistical significant difference between group I and group C for number of attempt for ventilating bougie insertion; Test type: Other; p > 0.05, Chi-squared, Corrected; Risk Ratio (RR) = 0.8972, 95% CI 2-sided [0.4858 to 1.6569]

3. Primary Outcome: Number of Attempts for Railroading of Endotracheal Tube Over Ventilating Bougie
Time Frame: 30 seconds
Measure: Number; unit: attempt
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
attempt
  1st attempt | 29 | 28
  2nd attempt | 0 | 1
  3rd attempt | 0 | 0
Statistical Analysis 1: Comparison: Group-I vs Group-C; Test type: Other; p > 0.05, Chi-squared, Corrected

4. Secondary Outcome: Heart Rate
Description: Heart rate to observe at the following time intervals.
  1. Base line
  2. After induction
  3. After dexmedetomidine injection
  4. Supraglottic airway insertion
  5. Ventilating bougie insertion
  6. ETT insertion
  7. 3minute after ETT insertion
  8. 5 minute after ETT insertion
  9. 7 minute after ETT insertion
  10. 10 minute after ETT insertion
  11. 15 minute after ETT insertion Study period is upto 15 minutes, thereafter the study ends here.
Time Frame: 25 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
beats per minute
  Baseline | 91.06 (11.72) | 88.89 (9.76)
  After Dex injection | 71.24 (9.98) | 72.75 (10.76)
  After induction | 69.87 (11.81) | 74.1 (11.17)
  SGA insertion | 75.68 (9.41) | 78.79 (9.73)
  V. Bougie insertion | 85.55 (6.60) | 82.41 (5.78)
  ETT insertion | 83.27 (9.75) | 81.65 (5.94)
  3 min after ETT insertion | 83.75 (8.78) | 82.72 (7.65)
  5 min after ETT insertion | 81.17 (6.99) | 79 (8.62)
  7 min after ETT insertion | 81.86 (7.01) | 79.34 (7.31)
  10 min after ETT insertion | 80.86 (6.53) | 78.79 (6.39)
  15 min after ETT insertion | 81.13 (5.87) | 78.41 (8.02)
Statistical Analysis 1: Comparison: Group-I vs Group-C; Heart rate beats per minute measured at base line among the group I and group C; Test type: Other; p = 0.44, t-test, 2 sided
Statistical Analysis 2: Comparison: Group-I vs Group-C; Heart rate beats per minute is measured following Dexmedetomidine injection among the group I and group C; Test type: Other; p = 0.58, t-test, 2 sided
Statistical Analysis 3: Comparison: Group-I vs Group-C; Heart rate beats per minute measured following induction of anaesthesia among the group I and group C; Test type: Other; p = 0.16, t-test, 2 sided
Statistical Analysis 4: Comparison: Group-I vs Group-C; Heart rate beats per minute measured following supraglottic airway insertion among the group I and group C; Test type: Other; p = 0.22, t-test, 2 sided
Statistical Analysis 5: Comparison: Group-I vs Group-C; Heart rate beats per minute measured following ventilating bougie insertion among the group I and group C; Test type: Other; p = 0.059, t-test, 2 sided
Statistical Analysis 6: Comparison: Group-I vs Group-C; Heart rate beats per minute measured at endotracheal intubation among the group I and group C; Test type: Other; p > 0.33, t-test, 2 sided
Statistical Analysis 7: Comparison: Group-I vs Group-C; Heart rate beats per minute measured after 3 minute of ETT insertion among the group I and group C; Test type: Other; p = 0.63, t-test, 2 sided
Statistical Analysis 8: Comparison: Group-I vs Group-C; Heart rate beats per minute measured after 5 minute of ETT insertion among the group I and group C; Test type: Other; p = 0.29, t-test, 2 sided
Statistical Analysis 9: Comparison: Group-I vs Group-C; Heart rate beats per minute measured after 7 minute of ETT insertion among the group I and group C; Test type: Other; p = 0.18, t-test, 2 sided
Statistical Analysis 10: Comparison: Group-I vs Group-C; Heart rate beats per minute measured after 10 minute of ETT insertion among the group I and group C; Test type: Other; p = 0.98, t-test, 2 sided
Statistical Analysis 11: Comparison: Group-I vs Group-C; Heart rate beats per minute measured after 15 minute of ETT insertion among the group I and group C; Test type: Other; p = 0.49, t-test, 2 sided

5. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure measured at following time intervals.
  1. Base line
  2. After Dexmedetomidine injection
  3. After induction of anaesthesia
  4. Supraglottic airway insertion
  5. Ventilating bougie insertion
  6. ETT insertion
  7. 3 minute after ETT insertion
  8. 5 minute after ETT insertion
  9. 7 minute after ETT insertion
  10. 10 minute after ETT insertion
  11. 15 minute after ETT insertion. The study period was upto 15 minutes and thereafter the study ends.
Time Frame: 25 minutes
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
mmhg
  Baseline | 122.31 (8.07) | 125.31 (11.06)
  After Dex injection | 109.96 (8.15) | 114.34 (12.41)
  After induction | 108.03 (8.34) | 112.51 (10.53)
  SGA insertion | 113.93 (6.14) | 114.24 (6.62)
  V. Bougie insertion | 118.65 (5.17) | 116.10 (4.73)
  ETT insertion | 117.37 (4.87) | 117.93 (6.70)
  3 min after ETT insertion | 116.03 (4.91) | 118.31 (8.1)
  5 min after ETT insertion | 118.62 (5.36) | 118.31 (8.1)
  7 min after ETT insertion | 115.13 (5.35) | 115.79 (6.95)
  10 min after ETT insertion | 116.93 (6.55) | 116.96 (10.95)
  15 min after ETT insertion | 116.62 (6.61) | 118.1 (9.54)
Statistical Analysis 1: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared at base line between group I and group C; Test type: Other; p = 0.24, t-test, 2 sided
Statistical Analysis 2: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared following Dexmedetomidine injection between group I and group C; Test type: Other; p = 0.11, t-test, 2 sided
Statistical Analysis 3: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared following induction os anaesthesia between group I and group C; Test type: Other; p = 0.07, t-test, 2 sided
Statistical Analysis 4: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared following supraglottic airway insertion between group I and group C; Test type: Other; p = 0.85, t-test, 2 sided
Statistical Analysis 5: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared following ventilating bougie insertion between group I and group C; Test type: Other; p = 0.055, t-test, 2 sided
Statistical Analysis 6: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared at ETT insertion time between group I and group C; Test type: Other; p = 0.71, t-test, 2 sided
Statistical Analysis 7: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared 3 minutes after ETT insertion between group I and group C; Test type: Other; p = 0.20, t-test, 2 sided
Statistical Analysis 8: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared 5 minutes after ETT insertion between group I and group C; Test type: Other; p = 0.86, t-test, 2 sided
Statistical Analysis 9: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared 7 minutes after ETT insertion between group I and group C; Test type: Other; p = 0.68, t-test, 2 sided
Statistical Analysis 10: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared 10 minutes after ETT insertion between group I and group C; Test type: Other; p = 0.98, t-test, 2 sided
Statistical Analysis 11: Comparison: Group-I vs Group-C; Systolic blood pressure measured and compared 15 minutes after ETT insertion between group I and group C; Test type: Other; p = 0.49, t-test, 2 sided

6. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure measured at following time intervals.
  1. Base line
  2. After Dexmedetomidine injection
  3. After Induction
  4. Supraglottic airway insertion
  5. Ventilating bougie insertion
  6. ETT insertion
  7. 3 minute after ETT insertion
  8. 5 minute after ETT insertion
  9. 7 minute after ETT insertion
  10. 10 minutes after ETT insertion
  11. 15 minute after ETT insertion The study period was upto 15 minutes. thereafter study ends.
Time Frame: 25 minutes
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
mmhg
  Baseline | 79.96 (5.88) | 81.51 (6.57)
  After Dex injection | 71.24 (7.67) | 73.68 (9.03)
  After induction | 70.1 (7.99) | 72.79 (8.64)
  SGA insertion | 75.24 (5.13) | 75.17 (8.37)
  V. Bougie insertion | 77.03 (4.22) | 76.51 (6.40)
  ETT insertion | 76.51 (5.19) | 75.68 (5.50)
  3 min after ETT insertion | 76.24 (4.04) | 75.34 (5.72)
  5 min after ETT insertion | 76.03 (4.38) | 75.03 (6.57)
  7 min after ETT insertion | 76.1 (4.38) | 75.72 (5.22)
  10 min after ETT insertion | 77.37 (3.60) | 76.79 (6.96)
  15 min after ETT insertion | 77.1 (4.35) | 76.79 (5.48)
Statistical Analysis 1: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared at base line between group I and group C; Test type: Other; p = 0.34, t-test, 2 sided
Statistical Analysis 2: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared following Dexmedetomidine injection between group I and group C; Test type: Other; p = 0.27, t-test, 2 sided
Statistical Analysis 3: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared following induction of anaesrthesia between group I and group C; Test type: Other; p = 0.22, t-test, 2 sided
Statistical Analysis 4: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared following supraglottic airway insertion between group I and group C; Test type: Other; p = 0.96, t-test, 2 sided
Statistical Analysis 5: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared following ventilating bougie insertion between group I and group C; Test type: Other; p = 0.71, t-test, 2 sided
Statistical Analysis 6: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared the time of endotracheal tube insertion between group I and group C; Test type: Other; p = 0.55, t-test, 2 sided
Statistical Analysis 7: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared 3 minutes after endotracheal tube insertion between group I and group C; Test type: Other; p = 0.49, t-test, 2 sided
Statistical Analysis 8: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared 5 minutes after endotracheal tube insertion between group I and group C; Test type: Other; p = 0.49, t-test, 2 sided
Statistical Analysis 9: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared 7 minutes after endotracheal tube insertion between group I and group C; Test type: Other; p = 0.76, t-test, 2 sided
Statistical Analysis 10: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared 10 minutes after endotracheal tube insertion between group I and group C; Test type: Other; p = 0.69, t-test, 2 sided
Statistical Analysis 11: Comparison: Group-I vs Group-C; Diastolic blood pressure measured and compared 15 minutes after endotracheal tube insertion between group I and group C; Test type: Other; p = 0.81, t-test, 2 sided

7. Primary Outcome: Time of Insertion
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
Seconds
  Supraglottic airway | 26.17 (2.25) | 44.65 (9.14)
  Ventilating bougie | 31.51 (8.87) | 26.31 (9.25)
  ETT | 25.58 (4.01) | 28.13 (8.31)
Statistical Analysis 1: Comparison: Group-I vs Group-C; We had compared time of insertion for supraglottic airway between group I and group C; Test type: Other; p < 0.0001, t-test, 2 sided

8. Primary Outcome: Total Intubation Time
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Group-I | Group-C
Number analyzed (Participants) | 29 | 29
Second | 93.27 (9.03) | 108.96 (16.50)
Statistical Analysis 1: Comparison: Group-I vs Group-C; Test type: Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Group-I | Group-C
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 2/29 | 4/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-I (N=29) | Group-C (N=29)
Airway trauma (Surgical and medical procedures) | 2 (2) | 3 (3) — Trauma to tongue, lips, teeth, pharyngeal tissue etc.
Tube impingement (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The use of fiber optic bronchoscope for confirmation of proper placement of I-gel and C-LMA would have been better. Also One can see the passage of ventilating bougie through I-gel and C-LMA into larynx and trachea.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No